CLINICAL TRIAL: NCT03174210
Title: Effects of Supplemental Oxygen Delivered by a Portable Oxygen Concentrator Compared to a Liquid Oxygen Device in Hypoxemic COPD Patients at Rest
Brief Title: Effects of Supplemental Oxygen Delivered by a Portable Oxygen Concentrator Compared to a Liquid Oxygen Device in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ActivoxTitration
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; supplemental oxygen; oxygen concentrator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: patients will be randomized into two different Groups (prospective cross-over design)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patients with delivery order 1, 2 (Experimental): Patients will use two different Oxygen devices at rest (1.liquid oxygen device (Companion R), 2. portable Oxygen concentrator (Activox TM 4L))
  Interventions: Device: liquid oxygen device (LOD); Device: portable oxygen concentrator (POC)
- COPD patients with delivery order 2,1 (Experimental): Patients will use two different Oxygen devices at rest (1. portable Oxygen concentrator (Activox TM 4L), 2. liquid oxygen device (Companion R))
  Interventions: Device: liquid oxygen device (LOD); Device: portable oxygen concentrator (POC)

INTERVENTIONS:
Device: liquid oxygen device (LOD) — This oxygen Supplementation is used in special order
  Other Names: Companion 1000 Chart Industries, Inc. Garfield Heights, USA
Device: portable oxygen concentrator (POC) — This oxygen Supplementation is used in special order
  Other Names: Activox™ 4L, Inovalabs Inc., Texas, USA

SUMMARY:
The aim of this study is to investigate the effects of supplemental oxygen on blood oxygenation at rest in Patients with severe to very severe COPD comparing the portable oxygen concentrator (Activox™ 4L) to a liquid continuous oxygen device (Companion®).

DETAILED DESCRIPTION:
It has been proven that supplemental oxygen increases oxygen saturation and reduces dyspnea in hypoxemic COPD Patients. There are different oxygen delivery systems available, some of them operating with liquid oxygen and others by concentrating the ambient air (concentrators). An advantage of the concentrator system is, that there is no refill required, but only a power plug and plug socket, enabling the patient for higher mobility and to be more autonomous. There are only few publications about whether portable oxygen concentrators have a comparable efficiency on oxygen saturation to liquid oxygen devices with continuous flow (LOD) or not. Until now there are no official recommendations about how to convert the oxygen flow rate for LOD (liter per minute) into the corresponding level of the POC.

Therefore, we investigate the comparability of the portable oxygen concentrator Activox™ 4L (POC) to a liquid oxygen device (Companion®) in 30 hypoxemic COPD patients at rest.

As a baseline assessment, the patients will receive a bodyplethysmography, blood gas analysis without using supplemental oxygen and an evaluation of the diffusion capacity of the lung for CO.

The study will be conducted on 2 consecutive days. 15 patients will be randomized into two different groups: First group will start with POC and will continue the following day with LOD; The second group will start with LOD and continue with POC (cross-over design). All patients will use the same oxygen devices during the study assessments (LOD: Companion 1000 (CE 0050), Chart Industries Inc., Garfiel Heights, OH, USA; POC: Activox™ 4L, Inovalabs Inc., Texas, USA). On both days of the study, patients will be connected to one of the two systems via nasal cannula for a total time period of 40 minutes, while the patient remains in a sitting position without talking. The oxygen flow rate starts at 1liter/min (LOD) or Level 1 (POC) and will be increased every 10 minutes to the next higher level until the maximum of 4l/min (LOD) or level 4 (POC) is reached. Blood gases were taken and breathing frequency will be recorded at the end of each Oxygen Level.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with hypoxemia at rest (paO2 < 55 or 60 mmHg, according to the recent supplemental oxygen guidelines [Hadringe, M., et al., British Thoracic Society guidelines for home oxygen use in adults. Thorax, 2015. 70 Suppl 1: p. i1-43.]
* Participation in an inpatient pulmonary rehabilitation program (Schön Klinik BGL)
* Written informed consent

Exclusion Criteria:

* The Need of more than 4 Liter/min Oxygen at rest to achieve PaO2 > 55 or 60mmHg
* Signs of acute exacerbation
* General exclusion criteria for exercise tests, e.g. acute coronary syndrome, acute myo- or pericarditis, acute lung embolism, pulmonary infarction, acute uncontrolled heart insufficiency

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Difference between LOD and POC in Partial pressure of oxygen levels | after 10 minutes of each LOD step compared to 10 minutes of each POC step
  PO2 values between LOD and POC at comparable Levels of oxygen supply (1liter/minute LOD will be compared to Level 1 of POC until 4liters/Minute LOD to Level 4 of POC)

SECONDARY OUTCOMES:
Difference between LOD and POC in Partial pressure of carbon dioxide levels | after 10 minutes of each LOD step compared to 10 minutes of each POC step
  PCO2 values between LOD and POC at comparable Levels of oxygen supply (1liter/minute LOD will be compared to Level 1 of POC until 4liters/Minute LOD to Level 4 of POC)
Change of partial pressure of Oxygen from one POC step to the next step | after 10 minutes of one POC step compared to after 10 minutes of the next POC step
  Change in PO2 values from e.g. POC step 1 to POC step 2, step 2 to 3 etc.
Change of partial pressure of carbon dioxide from one POC step to the next step | after 10 minutes of one POC step compared to after 10 minutes of the next POC step
  Change in PCO2 values between e.g. POC step 1 to POC step 2, step 2 to 3 etc.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof., Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Undecided